CLINICAL TRIAL: NCT01504997
Title: A Phase II Study of Robot Assisted Distal Gastrectomy With Nodal Dissection for Clinical Stage Ia Gastric Cancer
Brief Title: Phase II Study for Robot Assisted Distal Gastrectomy
Acronym: RADGphaseII
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shizuoka Cancer Center (Other)
Responsible Party: Principal Investigator, Masanori Terashima, Head of Gastric Surgery, Shizuoka Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DaVinci_SCC; UMIN000006910 (Other: UMIN)
Record Dates: First submitted 2011-12-30; First posted 2012-01-06 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Early Gastric Cancer
Keywords: DaVinci; Robot assisted surgery; Gastrectomy; Safety; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Robot assisted distal gastrectomy (Experimental): patients who received robot assisted distal gastrectomy
  Interventions: Device: Robot assisted distal gastrectomy (DaVinci)

INTERVENTIONS:
Device: Robot assisted distal gastrectomy (DaVinci) — patients who received robot assisted distal gastrectomy
  Other Names: DaVinci

SUMMARY:
The aim of this study is to clarify safety of robot assisted distal gastrectomy with lymph node dissection in patients with stage Ia early gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy specimen from the primary lesion shows adenocarcinoma
2. Diagnosed as Stage IA early gastric cancer according to the preoperative esophagogastroduodenoscopy and computer tomography
3. Endoscopic submucosal dissection is not indicated
4. Tumor was located within lower two thirds of stomach
5. Not having duodenal invasion
6. Eastern clinical oncology group performance status is 0 or 1
7. Body mass index is lower than 30
8. No prior laparotomy
9. No prior chemotherapy or radiation including those for other cancers
10. Fulfil all following conditions WBC > 3,000/mm3 Plt > 100,000/mm3 AST < 100 IU/L ALT < 100IU/L T.Bil < 2.0 g/dl Cre < 1.5mg/dl

Exclusion Criteria:

1. Having other active cancers
2. Possibly pregnant, or breast feeding woman
3. with psychiatric disorder
4. Receiving steroids
5. With Acute myocardial infarction in 6 months or with unstable angina
6. With uncontrolled hypertension
7. With uncontrolled diabetes mellitus
8. With pulmonary disease which require continuous oxygen therapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2017-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Masanori Terashima, M.D., Ph.D., Principal Investigator — Division of Gastric Surgery, Shizuoka Cancer Center
Locations (1):
- Shizuoka Cancer Center, Shizuoka, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 23 patients were recruited for the study, and the initial 5 cases were excluded from the primary analysis because some of the initial RAGs were performed by invited surgeons who had lots of experience. This exclusion was prespecified in the protocol. Therefore, only the remaining 18 patients were included in the analysis.
Period: Overall Study
Arm/Group | Robot Assisted Distal Gastrectomy
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Robot Assisted Distal Gastrectomy
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 65.5 [53 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Region of Enrollment [Number; unit: participants]
  Japan | 18

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Post-operative Intra-abdominal Infectious Complications
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 days
Measure: Number (90% Confidence Interval); unit: participants
Arm/Group | Robot Assisted Distal Gastrectomy
Number analyzed (Participants) | 18
participants | 0 [0 to 12]

2. Secondary Outcome: Overall Survival
Time Frame: 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Relapse Free Survival
Time Frame: 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Completion Rate of Robot Assisted Surgery
Time Frame: During the surgery, an expected average of 5 hours
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Adverse Events
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Robot Assisted Distal Gastrectomy
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes